CLINICAL TRIAL: NCT07330336
Title: 5-Year Follow-up of Children and Mother After Expectant Management Versus Induction of Labor in Low-risk Nulliparous Women at 39 Weeks of Gestation
Acronym: FAMILY-FA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: French Ministry of Social Affairs and Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2024/46
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Neurodevelopmental Disorders
Keywords: Child neurodevelopmental disorder; pregnancy; Low-risk nulliparous women; induction of labor; elective; cesarean delivery; maternal mental health; postpartum; depression
MeSH Terms: conditions — Neurodevelopmental Disorders; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- elective induction arm (Experimental): elective induction
  Interventions: Behavioral: Questionnaires
- expectant management arm (Active Comparator): expectant management
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — self-administered parental and teacher questionnaires 5 years after the birth of the first child (i.e., 5 years after enrollment in the FRENCH-ARRIVE trial). In addition, for a randomly selected subsample of 12% of participants (n=500), a brief neuropsychological assessment of their child (~1 hour) will be conducted remotely via videoconference by a trained neuropsychologist

SUMMARY:
In France, the rate of labor induction has markedly increased in recent years, partly following the ARRIVE trial suggesting short-term benefits of elective induction at 39 weeks in low-risk nulliparous women. This trial is currently being replicated in France (FRENCH-ARRIVE), as maternal characteristics, cesarean rates, and healthcare organization differ from the US. Importantly, no comparative data exist on the mid-term consequences of reducing gestational age at delivery with elective induction of labor-from 41 to 39 weeks-versus usual expectant management on child health and maternal outcomes. Generating such evidence is essential to inform decision making for women reaching 39 weeks of gestation, i.e. the large majority of pregnant women

DETAILED DESCRIPTION:
In France, the rate of labor induction increased from 20% to 25% of deliveries between 2016 and 2021. This recently dramatic increase also reported in other high income settings, is likely in part related to the publication of the ARRIVE trial (Grobman, NEJM 2018). Before it, induction of labor was usually proposed in case of condition potentially associated to a higher maternal or fetal risk with expectant management compared with an immediate delivery. The ARRIVE trial, a multicenter, randomized, controlled trial suggests a short-term maternal-fetal benefit to systematic induction of labor at 39 weeks of gestation (experimental arm) compared to an expectant management (control arm) in low-risk nulliparous women, with a decreasing trend of adverse perinatal outcome and a significant lower risk of cesarean delivery and maternal hypertensive disorders. Because the generalizability of these results in US outside settings is unknown (as the maternal characteristics, national rate of cesareans and organization and access of care differ in US from an European country including France, this trial is currently replicating in France (FRENCH-ARRIVE trial, PHRCN n° 19-0063) (Sentilhes et al, Lancet 2023; Azria et al, AJOG 2023;)

Regardless of its results (which are not yet available), mid-term follow-up of children born to mothers enrolled in the FRENCH-ARRIVE trial, through the FAMILY-FA project, is crucial:

1 / In absence of comparative data, it remains unknown whether the mid-term child health differs or not according to the late pregnancy management, through the bias of reduction the gestational age at delivery from 41 to 39 weeks for women undergoing an induction of labor, and with possible differences in mode of delivery (all these parameters being associated to mid-term child's health).

2/ For the informed decision making for the women who reach 39 weeks gestation (i.e. the large majority of the pregnant women). Only mid-term data in early childhood after induction of labor for medical reason compared to expectant management are available; but they are obviously flawed by the indication that required the induction of labor (e.g. fetal growth restriction, premature of membranes, etc).

Thus, the first objective of the FAMILY-FA project is to evaluate the mid-term effect of elective induction of labor at 39 weeks of gestation compared with an expectant attitude in low-risk nulliparous women on child neurodevelopment at 5 years.

Similarly, mid-term follow-up of mothers enrolled in the FRENCH-ARRIVE trial with the assessment of obstetrical issues in case of future pregnancy, and maternal mental health, through the FAMILY-FA project, is essential:

1. No comparative data are available on the obstetrical issues including mode of delivery in case of a subsequent pregnancy (the possible reduction of cesarean associated to the elective induction of labor at 39 weeks compared to an expectant management might be associated to a lower rate of cesarean and maternal and neonatal morbidity in a subsequent pregnancy).
2. We have recently shown that induction of labor for medical reason was associated with impairment of maternal mental health in postpartum
3. By assessing the maternal mental health as well as the other components of the life of the women (single or not, subsequent pregnancy or not) concomitantly to assessing the offspring development will allow us to taking into account potential cofounders associated to pediatric neurodevelopment (primary objective of our project). In fact, high quality evidence show that impaired maternal mental health affects intra-familial relationships and may impair the child's development.

ELIGIBILITY:
Inclusion Criteria:

* Women randomized in the FRENCH-ARRIVE trial (NCT04799912):

  * Age ≥ 18 years
  * Nulliparous women (i.e. no previous pregnancy beyond 20 weeks)
  * With singleton gestation. Twin gestation reduced to singleton, either spontaneously or therapeutically, is not eligible unless the reduction occurred before 14 weeks project gestational age.
  * Gestational age at randomization between 37 weeks of gestation 0 day and 38 weeks of gestation 6 days inclusive based on the crown rump length measured at the first trimester ultrasound before 14 weeks of gestation and 0 days, as recommended in France
  * Affiliated or beneficiary to a health security system
  * Signed informed consent
* Non-opposition from both holders of parental authority to participation in the FAMILY-FA study

Exclusion Criteria:

* Exclusion criteria of the FRENCH-ARRIVE trial:

  * Project gestational age at date of first ultrasound is > 14 weeks
  * Plan for induction of labor prior to 40 weeks 5 days
  * Plan for cesarean delivery or contraindication to labor
  * Breech presentation
  * Multiple pregnancy
  * Signs of labor (regular painful contractions with cervical change)
  * Fetal demise or known major fetal anomaly
  * Heparin or low-molecular weight heparin during the current pregnancy
  * Placenta previa, accreta, vasa previa
  * Active vaginal bleeding greater than bloody show
  * Ruptured membranes
  * Cerclage in current pregnancy
  * Known oligohydramnios, defined as Amniotic Fluid Index < 5 or Maximal Vertical Pocket < 2 cm
  * Fetal growth restriction, defined as Estimated Fetal Weight < 10th percentile according to local curve
  * Known HIV positivity because of modified delivery plan
  * Major maternal medical illness associated with increased risk for adverse pregnancy outcome (for example, any diabetes mellitus, lupus, any hypertensive disorder, cardiac disease, renal insufficiency)
  * Refusal of blood products
  * Participation in another interventional study that may influence management of labor or delivery (labor induction, operative vaginal delivery, cesarean section, shoulder dystocia)
  * Delivery planned elsewhere at a non-Network site
  * History of myomectomy by laparotomy or laparoscopy
  * Previous metroplasty for uterine malformation or Asherman syndrome
  * Patient under legal protection
  * Poor understanding of the French language
* Moreover: the following postnatal criteria will be also exclusion criteria:

  * Major malformations and/or chromosomal aberrations evidenced in the child after birth
  * Parents' refusal to participate in the follow-up
  * Impossibility to contact the family

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4200 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2032-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
pediatric neurodevelopment at 5 years of age | 5 years old
  pediatric neurodevelopment at 5 years of age, based on the assessment of different dimensions (development, motor, coordination, neurosensory, language, and behavior and executive functions). The Ages and Stages Questionnaire (ASQ-3) and the preschool version of the Child Behavior Checklist (CBCL 1½-5). The scales will be analyzed quantitatively, and the extreme values of the scores obtained will be considered pathological (≥2SD below mean or <83th percentile, depending on the scale) according to the literature

SECONDARY OUTCOMES:
Child neurodevelopment | 5 years old
  Neurodevelopment at 5 years of age, based on the Global School Adaptation score (GSA score) which has been shown to have a good correlation to cognitive abilities (see below) (4): Six questions investigate linguistic competence and 5 questions investigate non-verbal abilities. Eight questions address children's behavior in the classroom. The final question invites the teacher to give his or her prognosis for the child's future adaptation to school life. A score over 45 was defined as a positive evaluation of the child's adaptation to school life.
Child cognition | 5 years old
  Cognition (intellectual ability), evaluated using the WPPSI-IV (Wechsler Preschool & Primary Scale of Intelligence), which measures cognitive ability in five domains (verbal comprehension, visuospatial indices, fluid reasoning, working memory, processing speed) resulting in a composite full scale intelligence quotient reflecting the overall level of intelligence. The test will be based on an online neuropsychological assessment for a random sample of 12% (N=500) of mother included in the FRENCH-ARRIVE trial
Maternal depression | Baseline
  Maternal mental health including depression evaluated using the Beck Depression Inventory (BDI-II), a 21-item self-reported rating inventory that measures attitudes and symptoms of depression and screens for self-harm. The BDI-II score ranges from 0 to 63. A score of 0 to 13 suggests minimal depression; 14 to 19, mild depression; 20 to 28, moderate depression; and 29 to 63, severe depression
Maternal anxiety | Baseline
  Maternal mental health including anxiety evaluated using the 7-item Generalized Anxiety Disorder Questionnaire (GAD-7) measuring anxiety severity and which contains 7 items scored on a 0- to 3-point scale, with higher scores indicating worse anxiety. The GAD-7 has been validated in postpartum samples. A difference of 4 points defined a clinically significant change
Maternal partner relationship satisfaction | Baseline
  Partner relationship satisfaction assessed via maternal report on the 5-item short version Relationship Satisfaction Scale (RSS). Items were rated on a 6-point scale to reflect relationship satisfaction (eg, "I am very happy with our relationship") and partner relationship quality (eg, "my partner is generally understanding"). The scale consists of 10 statements to be answered on a 6-point scale from 1-strongly disagree to 6-strongly agree. Total scores range from 10 to 60, with lower scores indicating less satisfaction with the relationship.
Maternal precarity | Baseline
  Precarity, assessed using the EPICES score (Evaluation de la Précarité et des Inégalités de santé dans les Centres d'Examens de Santé), an individual indicator of precarity that takes into account the multidimensional nature of precarity. The score is continuous, ranging from 0 (no precarity) to 100 (maximum precarity). The threshold of 30 is considered to be the precarity threshold according to EPICES working group.
Maternal life questionnaire | Baseline
  Life questionnaire, assessed using simple questions asking the patient about her family status (e.g. "Are you in a relationship?"; "Are you in a relationship with the co-parent of your first child?"), and previous psychiatric history (e.g. "Have you ever consulted a psychiatrist ?"; "Have you ever consulted a psychologist?"; "Did you experience depression the year after the birth of your first child?"; "Have you ever taken psychotropic drugs?"). These simple questions are essential to gather information on any psychosocial comorbidities that may be confounding factors in the assessment of the child at age 5

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France